CLINICAL TRIAL: NCT05952427
Title: Adverse Childhood Experiences and Infertility : ACESI
Acronym: ACESI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-A00776-39
Record Dates: First submitted 2023-06-26; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-06

CONDITIONS: Infertility, Female; Trauma, Psychological; Child Development; Child Abuse; Health Behavior
Keywords: psychologic; traumatism; women; sterility; infertility; abuse; development; gynecologist
MeSH Terms: conditions — Infertility, Female; Psychological Trauma; Health Behavior; Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infertile women: Any patient consulting for the first time at the Grenoble University Hospital in a context of infertility, between 18 and 43 years old
  Interventions: Other: ACE Questionnaire
- Non-infertile women: Any patient consulting her gynecologist in town for a reason other than infertility, and having no known infertility, between 18 and 43 years old
  Interventions: Other: ACE Questionnaire

INTERVENTIONS:
Other: ACE Questionnaire — The only intervention consists of completing the validated ACE questionnaire

SUMMARY:
Adverse childhood experiences can have powerful effects on health and quality of life in adulthood. Thus, having a history of childhood trauma, before the age of 18 (physical aggression, sexual abuse, death of a close person, etc.) significantly increases the risk of having cancer, cardiovascular disease, psychological damage , or earlier mortality. Validated scores allow the evaluation of the importance of adverse childhood experiences, in particular the ACE score (adverse childhood experiences) published by Felitti. Studies on the subject show a dose-response relationship between exposure to adverse childhood experiences and negative outcomes in terms of health and well-being. The physiopathological tracks to explain the occurrence of somatic pathologies in adulthood include the observation of a state of hyper-activation of the HPA axis that persists in adulthood; modulations of immunity, but also epigenetic modifications. Some data are available on the associations between childhood trauma and obstetric risks, with a significant increase in the risk of preterm delivery and fetal death in utero.

Primary objective :

1a) To study the prevalence of adverse childhood experiences (ACE) in women consulting for the first time in an PMA service for the desire to become pregnant, and 1b) To study the association between adverse childhood experiences and infertility in adulthood, by comparing infertile women with nulliparous control women in the general population consulting for their classic gynecological follow-up.

DETAILED DESCRIPTION:
Procedures for recruiting participants:

Cases (infertile women): A poster presenting the study will be put up in the waiting room of the PMA center of the Grenoble University Hospital. The information and non-objection letter as well as the ACE questionnaire will be made available to them in the waiting room. If the patient agrees to participate, she will complete the questionnaire completely anonymously and submit it to the secretariat.

Witnesses: A poster presenting the study will be put up in gynecology practices (Non-exhaustive list: Cabinet Gynelac of Dr Flandrin in Aix les Bains, Cabinet of Dr Chabre Groupe Hospitalier Mutualiste in Grenoble, Cabinet of Dr Fragai in Voiron , Cabinet of Dr. Biot at the Clinique des Cèdres in Echirolles, etc.) thus any woman consulting for a gynecological follow-up will be able to find out about the study.

The information and non-objection letter as well as the ACE questionnaire will be made available to them in the waiting room. If the patient agrees to participate, she will complete the questionnaire completely anonymously and submit it to the secretariat.

After inclusion, case women and control women will benefit from the usual care in the PMA center, or by their usual gynecologist. The participation of subjects in this study will in no way modify their care. The participation of the subjects will be limited to filling out the ACE questionnaire. No additional visit, no sampling or additional treatment other than those commonly carried out for the care of infertile women is carried out for this study.

If after answering the questionnaire, patients feel the need, they can be directed to the "Maison Des Femmes" in Grenoble, where they can benefit from appropriate multidisciplinary care (doctors, psychologists, physiotherapists, etc.).

Modalities of information and traceability of the non-opposition:

Cases (infertile women): the information letter will be available in the waiting room. The questionnaire being anonymous, there will be no possibility of opposition after having answered the questionnaire.

Witnesses: the newsletter will be available in the waiting room. The questionnaire being anonymous, there will be no possibility of opposition after having answered the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

- Case: Infertile adult women, nulliparous, aged 18 to 43, consulting for the first time at the clinical-biological center of AMP of the CHU of Grenoble Alpes for desire of pregnancy within the framework of a heterosexual couple

. - Controls: Women of legal age, nulliparous, in the general population consulting their city gynecologist during the same study period, aged 18 to 43 and a priori without known infertility

Exclusion Criteria:

* Patients who do not speak French well enough to benefit from clear and intelligible information
* Patients refusing to participate in the study

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women only
Study Population: Infertile adult women, nulliparous, aged 18 to 43, consulting for the first time at the clinical-biological center of AMP of the CHU of Grenoble Alpes for desire of pregnancy within the framework of a heterosexual couple
  * Controls: Women of legal age, nulliparous, in the general population consulting their city gynecologist during the same study period, aged 18 to 43 and a priori without known infertility
  * Case: Infertile adult women, nulliparous, aged 18 to 43, consulting for the first time at the clinical-biological center of AMP of the CHU of Grenoble Alpes for desire of pregnancy within the framework of a heterosexual couple
Sampling Method: Non-Probability Sample
Enrollment: 332 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence estimated by the proportion of patients with a high Adverse Childhood Experiences (ACE) score defined by a score ≥ 4, with Odds ratio and its 95% CI | the 1 day of the inclusion, starting from the first of august 9:00 am
  Prevalence of adverse childhood experiences (ACE) in women consulting for the first time in a PMA service for pregnancy desire, compared to women in the general population

SECONDARY OUTCOMES:
Description of types of adverse experiences | the 1 day of the inclusion, starting from the first of august 9:00 am
  Description of unfavorable childhood experiences among women consulting for pregnancy in an PMA service, using a validated score: the ACE score (CDC, 2021; Felitti et al., 1998).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Felitti VJ, Anda RF, Nordenberg D, Williamson DF, Spitz AM, Edwards V, Koss MP, Marks JS. REPRINT OF: Relationship of Childhood Abuse and Household Dysfunction to Many of the Leading Causes of Death in Adults: The Adverse Childhood Experiences (ACE) Study. Am J Prev Med. 2019 Jun;56(6):774-786. doi: 10.1016/j.amepre.2019.04.001. PMID 31104722
- [Background] Chrousos GP, Torpy DJ, Gold PW. Interactions between the hypothalamic-pituitary-adrenal axis and the female reproductive system: clinical implications. Ann Intern Med. 1998 Aug 1;129(3):229-40. doi: 10.7326/0003-4819-129-3-199808010-00012. PMID 9696732
- [Background] Harris HR, Wieser F, Vitonis AF, Rich-Edwards J, Boynton-Jarrett R, Bertone-Johnson ER, Missmer SA. Early life abuse and risk of endometriosis. Hum Reprod. 2018 Sep 1;33(9):1657-1668. doi: 10.1093/humrep/dey248. PMID 30016439
- [Background] Liebermann C, Kohl Schwartz AS, Charpidou T, Geraedts K, Rauchfuss M, Wolfler M, von Orelli S, Haberlin F, Eberhard M, Imesch P, Imthurn B, Leeners B. Maltreatment during childhood: a risk factor for the development of endometriosis? Hum Reprod. 2018 Aug 1;33(8):1449-1458. doi: 10.1093/humrep/dey111. PMID 29947745
- [Background] Jacobs MB, Boynton-Jarrett RD, Harville EW. Adverse childhood event experiences, fertility difficulties and menstrual cycle characteristics. J Psychosom Obstet Gynaecol. 2015;36(2):46-57. doi: 10.3109/0167482X.2015.1026892. Epub 2015 Mar 31. PMID 25826282
- [Background] Schliep KC, Mumford SL, Johnstone EB, Peterson CM, Sharp HT, Stanford JB, Chen Z, Backonja U, Wallace ME, Buck Louis GM. Sexual and physical abuse and gynecologic disorders. Hum Reprod. 2016 Aug;31(8):1904-12. doi: 10.1093/humrep/dew153. Epub 2016 Jun 22. PMID 27334336